CLINICAL TRIAL: NCT05347758
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-7535 in Healthy Subjects
Brief Title: A Phase I Single- and Multiple- Ascending Dose and Food Effect Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-7535 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: HRS-7535-101
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: HRS-7535 tablet compared with placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Drug: HRS-7535
  Interventions: Drug: HRS-7535
- Group B (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-7535 — Drug: HRS-7535
  Arms: Group A
Drug: Placebo — Drug: Placebo
  Arms: Group B

SUMMARY:
This is a randomized, double-blinded, placebo-controlled study to evaluate the safety, tolerability, Pharmacokinetics and Pharmacodynamics of single ascending dose (Part A) and multiple ascending dose (Part B) of HRS-7535 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 to 55 years of age (inclusive) healthy male or female of nonchildbearing potential;
2. Body weight of at least 50 kg for male, and 45 kg for female; and Body Mass Index (BMI) within the range of 19 to 28 kg/m2 (inclusive);
3. Subjects (including partners) of childbearing potential are willing to use protocol specified effective methods of contraception from screening to at least 6 months after the final dose of study drug;
4. Able and willing to provide written informed consent and to comply with the study protocol;
5. Physical examination, vital signs are normal or are judged not clinically significant by the investigator;

Exclusion Criteria:

1. Participants with any abnormal results and judged clinically significant by the investigator;
2. HbA1c ≥6.2%, fasting blood-glucose ≤3.9mmol/L (70mg/dL) or ≥6.1mmol/L(110mg/dL) at screening ;
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2 x ULN; total bilirubin ≥1.5 x ULN at screening;
4. Abnormal ECG that is clinically significant, or QTcF >450 msec;
5. Positive test result of any of the following at screening: hepatitis B surface antigen (HBsAg), hepatitis C antibody, syphilis, or human immunodeficiency virus (HIV) antibody;
6. Any malignancy (except basal cell carcinoma and squamous cell carcinoma of the skin) in the previous 5 years;
7. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, history of pancreatitis or symptomatic gallbladder disease;
8. History of gastric emptying anomalies (gastric outlet obstruction), severe chronic gastrointestinal diseases (such as inflammatory bowel disease, active ulcer) ;
9. Subject with major medical history of heart, liver, kidney, endocrine, digestive, blood, respiratory and genitourinary system or existing diseases of the above systems;
10. Use any prescription drugs, non-prescription drugs, food supplements, vitamins and Chinese herbal medicines within 2 weeks before administration;
11. Subject who received bariatric surgery or procedures, or use of weight-reducing drugs within 3 months prior to administration, or body weight change of more than ±10% within 3 months prior to administration;
12. Use any drugs that may affect glucose metabolism were used within 1 month before administration.
13. Suspected allergy to any ingredient in the study drug;
14. Participation in clinical trials of any drug or medical device within 3 months before screening;
15. History of regular alcohol consumption exceeding 14 drinks per week within 6 months before screening;
16. More than 5 cigarettes per day or cigarettes within 3 months before screening;
17. Subjects who consume alcoholic beverages, Seville oranges, grapefruit or juices, or products containing caffeine or xanthine (such as coffee, tea, cola drinks and chocolate) from 2 days before the start of study treatment;
18. Strenuous exercise in 48 hours before treatment;
19. Subjects with a history of drug abuse, drug dependence, or a positive drugs of abuse test, or a positive alcohol breath test before study drug administration;
20. Donation or loss of blood of ≥ 200 mL within 1 month or of ≥ 400 mL within 3 months prior to the first dose of study drug;
21. Subjects can't tolerate venipuncture;
22. Subjects have special dietary requirements and cannot comply with the unified diet;
23. Other conditions judged by the investigator to be not suitable to participate in the trial;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-18 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of adverse Events | Day-2 to last follow-up
  Number of adverse events per subject, including clinically relevant changes in physical examination, vital signs, laboratory tests and ECGs;

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of HRS-7535 - AUC0-t | pre-dose to 96 hours post-dose
  Area under the concentration-time curve from time zero to the last quantifiable time point t (AUC0-t);
Pharmacokinetic (PK) profile of HRS-7535 - AUC0-∞ | pre-dose to 96 hours post-dose
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞);
Pharmacokinetic (PK) profile of HRS-7535 - Cmax | pre-dose to 96 hours post-dose
  Maximum observed concentration (Cmax);
Pharmacokinetic (PK) profile of HRS-7535 - Tmax | pre-dose to 96 hours post-dose
  Time to maximum observed concentration (Tmax);
Pharmacokinetic (PK) profile of HRS-7535 - t1/2 | pre-dose to 96 hours post-dose
  Terminal elimination half-life (t1/2)
Pharmacokinetic (PK) profile of HRS-7535 - CL/F | pre-dose to 96 hours post-dose
  Apparent clearance (CL/F);
Pharmacokinetic (PK) profile of HRS-7535 - Vz/F | pre-dose to 96 hours post-dose
  Apparent volume of distribution (Vz/F);
Pharmacokinetic (PK) profile of HRS-7535 - AUC0-τ,ss | pre-last dose to 96 hours post- last dose
  Area under the plasma concentration-time curve from time zero to tau at steady state (AUC0-τ,ss)
Pharmacokinetic (PK) profile of HRS-7535 - AUC0-t,ss | pre- last dose to 96 hours post- last dose
  AUC0-t at steady state (AUC0-t,ss)
Pharmacokinetic (PK) profile of HRS-7535 - AUC0-∞,ss | pre- last dose to 96 hours post- last dose
  AUC0-∞ at steady state (AUC0-∞,ss)
Pharmacokinetic (PK) profile of HRS-7535 - Tmax,ss | pre- last dose to 96 hours post- last dose
  Tmax at steady state (Tmax,ss)
Pharmacokinetic (PK) profile of HRS-7535 - Cmax,ss | pre- last doseto 96 hours post- last dose
  Cmax at steady state (Cmax,ss)
Pharmacokinetic (PK) profile of HRS-7535 - Ctrough,ss | pre- last dose to 96 hours post- last dose
  Ctrough at steady state (Ctrough,ss)
Pharmacokinetic (PK) profile of HRS-7535 - Cavg,ss | pre- last dose to 96 hours post- last dose
  Cavg at steady state (Cavg,ss)
Pharmacokinetic (PK) profile of HRS-7535 - DF | pre- last dose to 96 hours post- last dose
  Degree of fluctuation at steady state (DF)
Pharmacokinetic (PK) profile of HRS-7535 - Vz,ss/F | pre- last dose to 96 hours post- last dose
  Vz/F at steady state (Vz,ss/F)
Pharmacokinetic (PK) profile of HRS-7535 - CLss/F | pre- last dose to 96 hours post- last dose
  CL/F at steady state (CLss/F)
Pharmacokinetic (PK) profile of HRS-7535 - t1/2,ss | pre- last dose to 96 hours post- last dose
  t1/2 at steady state (t1/2,ss)
Pharmacodynamic (PD) profile of doses of HRS-7535 - blood glucose | pre-dose to 24 hours post-dose
Pharmacodynamic (PD) profile of doses of HRS-7535 - insulin | pre-dose to 24 hours post-dose
Pharmacodynamic (PD) profile of doses of HRS-7535 - C-peptide | pre-dose to 24 hours post-dose
Pharmacodynamic (PD) profile of doses of HRS-7535 - glucagon | pre-dose to 24 hours post-dose
Pharmacodynamic (PD) profile of doses of HRS-7535 - fructosamine | pre-dose up to 96 hours after the last dose
PD profile of multiple doses of HRS-7535 - HbA1c | pre-dose up to 96 hours after the last dose
PD profile of multiple doses of HRS-7535 - 5-points glucose profile | pre-dose up to 24 hours after the last dose
PD profile of multiple doses of HRS-7535 - weight | pre-dose up to 96 hours after the last dose

IPD SHARING:
Plan to Share IPD: Undecided